CLINICAL TRIAL: NCT04961944
Title: HypErsensitiVity PneumonITis: DiseAse Progression Characterization. An International Multicentric Prospective Observational Study
Brief Title: HypErsensitiVity PneumonITis: DiseAse Progression Characterization
Acronym: EVITA
Status: Recruiting | Type: Observational
Sponsor: Hospital do Coracao (Other)
Collaborators: Boehringer Ingelheim (Industry); Centro Rossi, Buenos Aires, Argentina (Unknown)
Responsible Party: Sponsor
Other Study IDs: EVITA BI 1199-0430
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Hypersensitivity Pneumonitis
Keywords: hypersensitivity pneumonitis; pulmonary fibrosis; interstitial lung disease
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic; Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Respiratory Physiological Phenomena; Blood Specimen Collection; Genome; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Genomic DNA from blood; Blood for protein biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypersensitivity pneumonitis: see elegibility criteria
  Interventions: Other: Disease assessment

INTERVENTIONS:
Other: Disease assessment — A comprehensive evaluation of the disease's extension, its impact on function, quality of life, and the search for phenotype/endotypes will be performed.
  The association between endotypes and disease progression will be tested.
  Other Names: Pulmonary function test (PFT); High Resolution Computed Tomography (HRCT) of the Chest; 6-minute walking distance (6MWD); blood for genomics, functional genomics and protein biomarker analysis; urine collection for protein biomarker analysis; Bronchoalveolar fluid collection (in a subset of the sample); K-BILD questionnaire

SUMMARY:
EVITA is a multicentric Latin-American prospective cohort on chronic hypersensitivity pneumonitis. EVITA's objective is to identify phenotypes and/or endotypes associated with different disease trajectories measured primarily by forced vital capacity (FVC) during a 24 month follow-up period. Other secondary measures of disease progression will also be investigated such as imaging, time to death or lung transplantation, and patient-reported outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatient subjects (18 years old or older) that fulfill the 2020 ATS/JRS/ALAT diagnostic criteria of HP of at least moderate confidence (70% confidence or more).
2. Willingness to undergo the evaluations proposed in this protocol
3. HP diagnosis within the last 24 months
4. Presence of radiological or histological fibrosis:

4.a. Radiological fibrosis consists of unequivocal fine or coarse reticulation with architectural lung distortion and/or traction bronchiectasis and/or honeycomb.

4.b. Unequivocal histopathological fibrosis evidenced on lung specimens

Exclusion Criteria:

1. Pregnancy
2. Presence of established connective tissue disease
3. Severe comorbidity impacting on the respiratory system as judged by the attending physician (ex. congestive heart failure, neoplasm, post-COVID-19 sequelae)
4. Use of supplemental oxygen at rest
5. Dyspnea mMRC 4 (too breathless to leave the house or breathless when dressing or undressing)
6. Unequivocal emphysematous pattern of HP on HRCT
7. Unequivocal pleuro-parenchymal fibroelastosis on the HRCT
8. Significant pulmonary arterial hypertension:

8.a. Signs of right ventricular failure by echodopplercardiogram or 8.b. Cardiac index < 2L/min/m2 or right heart catheterism

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic (fibrotic) hypersensitivity pneumonitis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Variation in Forced Vital Capacity (FVC) as a continuous variable | 24 months

SECONDARY OUTCOMES:
Variation in Computed Tomography Lung Densitometry | 24 months
Time to death or lung transplantation | 24 months
Acute exacerbation rate | 24 months
King´s Brief Interstitial Lung Disease Questionnaire (K-BILD) | 24 months

OTHER OUTCOMES:
Proportion of patients varying FVC >= 10% | 24 months
Variation in meters walked measured by the 6MWT | 24 months
Variation in the ratio dessaturation/meters-walked measured by 6MWT | 24 months
Variation in the dyspnea scores on mMRC scale | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Kawano Dourado, MD, Principal Investigator — HCOR Research Institute, Hospital do Coracao, São Paulo, Brazil; Prof. Alexandra Latini, PhD, Study Chair — Federal University of Santa Catarina
Locations (10):
- Argentina (3):
  - Hospital Prov de Tórax Dr. A. Cetrángolo, Bueno Aires
  - Instituto de Rehabilitacion Psicofisica, Buenos Aires
  - University of Buenos Aires, Buenos Aires
- Brazil (6):
  - LABOX - Federal University of Santa Catarina, Santa Catarina, Santa Catarina
  - LAPOGE - Federal University of Santa Catarina, Santa Catarina, Santa Catarina
  - University Hospital HU Professor Polydoro - Federal University of Santa Catarina, Florianópolis
  - Centro EDUMED, Paraná
  - Hospital do Servidor Estadual de Sao Paulo (IAMPSE), São Paulo
  - InCor - Medical School of the University of Sao Paulo, São Paulo
- Instituto Nacional del Tórax, Santiago, Chile

IPD SHARING:
Plan to Share IPD: Undecided